CLINICAL TRIAL: NCT04405544
Title: Determination of Acute Encephalopathy Predictors in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Oleg Vinogradov, MD, PhD, State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NMSC-01-20
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Encephalopathy; COVID
MeSH Terms: conditions — Brain Diseases | interventions — Tomography, X-Ray Computed; Electroencephalography; Oximetry; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main (Other): patients with COVID-19 and Acute Encephalopathy
  Interventions: Diagnostic Test: CT-scan; Diagnostic Test: EEG; Diagnostic Test: EP; Diagnostic Test: Pulse oximetry; Diagnostic Test: Blood tests
- Control (Other): patients with COVID-19 without Acute Encephalopathy
  Interventions: Diagnostic Test: CT-scan; Diagnostic Test: EEG; Diagnostic Test: EP; Diagnostic Test: Pulse oximetry; Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: CT-scan — chest CT-scan
Diagnostic Test: EEG — Electroencephalography
Diagnostic Test: EP — Evoked potential
Diagnostic Test: Pulse oximetry — Pulse oximetry
Diagnostic Test: Blood tests — Blood tests

SUMMARY:
The SARS-CoV-2 infection was detected in December 2019 in Wuhan City, China. The infection affects all age groups, although childhood is the lowest proportion of those affected.

The main clinical manifestations that require hospitalization of infected patients are SARS pneumonia, which may require treatment in the intensive care unit (27%) and its progression into acute respiratory distress syndrome (67%) with life-threatening conditions in almost 25% of patients diagnosed with "SARS-CoV-2 infection".

Nervous system damage with SARS-CoV-2 infection has been practically not investigated, but neurological disorders have been reported in 36% of these patients.

Finally, the mortality rate associated with the new virus is high in patients who require treatment in intensive care units (62% of cases).

Therefore, we are conducting a prospective study to identify acute encephalopathy predictors in patients with COVID-19.

DETAILED DESCRIPTION:
This is a prospective, cohort-based, adaptive design study that aims to identify acute encephalopathy predictors in patients with COVID-19. Patients with community-acquired pneumonia and confirmed pulmonary tissue infiltration will be enrolled in the study based on CT data with changes corresponding to the medium and high probability of coronavirus pneumonia (CO-RADS 4-5) and lesion of at least 25% of one lung.

Each patient will be examined at least twice (2 visits): P1 - on admission to hospital; P2 - in 10±5 days.

In the further course of the disease patients will be divided into 2 groups (cohorts). Group 1 - patients who have developed acute encephalopathy. Group 2 - patients who at the moment of discharge have no acute encephalopathy.

The study will collect clinical exam ( including neurological signs), neurophysiological data (including electroencephalography (EEG) and evoked potential (EP)), comprehensive laboratory tests, CT-scan and all standards of care to identify predictors of acute encephalopathy.

The study will consist of two phases:

1. The pilot phase - inclusion of the first 60 patients, followed by an interim analysis on the basis of which will be clarified:

   * sample size;
   * clinical, laboratory and instrumental parameters to be analyzed;
   * terms and frequency of the EEG and EP.
2. The main phase - further patient recruitment and all procedures required by the protocol.

The intermediate and final analysis will include both patients who have developed acute encephalopathy (main group) and patients who have not developed acute encephalopathy (control group).

Acute encephalopathy will be defined as recently stated :

1. The term acute encephalopathy refers to a rapidly developing (over less than 4 weeks, but usually within hours to a few days) pathobiological process in the brain. This is a preferred term
2. Acute encephalopathy can lead to a clinical presentation of subsyndromal delirium, delirium, or in case of a severely decreased level of consciousness, coma; all representing a change from baseline cognitive status
3. The term delirium refers to a clinical state characterized by a combination of features defined by diagnostic systems such as the DSM-5.

Delirium according to the DSM-5 is defined if criterium A-E are fulfilled:

A. Disturbance in attention (i.e., reduced ability to direct, focus, sustain, and shift attention) and awareness (reduced orientation to the environment).

B. The disturbance develops over a short period of time (usually hours to a few days) represents a change from baseline attention and awareness, and tends to fluctuate in severity during the course of the day.

C. An additional disturbance in cognition (e.g., memory deficit, disorientation, language, visuospatial ability, or perception).

D. The disturbances in criteria A and C are not explained by another pre-existing, established, or evolving neurocognitive disorder, and do not occur in the context of a severely reduced level of arousal, such as coma.

E. There is evidence from the history, physical examination, or laboratory findings that the disturbance is a direct physiologic consequence of another medical condition, substance intoxication or withdrawal (i.e. because of a drug of abuse medication), or exposure to a toxin, or is because of multiple etiologies [1].

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 60 years
* Out-of-hospital pneumonia with confirmed pulmonary tissue infiltration according to CT with changes corresponding to the average and high probability of coronavirus pneumonia (4-5 levels by CO-RADS classification) and the loss of more than 25% of one of the lungs.
* The patient has read the information sheet and signed the informed consent form.

Exclusion Criteria:

* Negative PCR test for coronavirus infection.
* The presence in the anamnesis of data for myocardial infarction or stroke.
* Verified thrombophilia.
* Pregnancy.
* Patients with malignant tumors (including anamnesis), including postoperative period in the background of chemo and/or radiation therapy.
* Acute stroke.

Dropout Criteria:

* Patient's refusal to participate further in the study.
* Negative PCR result for coronavirus infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who have developed encephalopathy | 10 days
  The percentage of patients who have developed encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Oleg I Vinogradov, MD, PhD, Principal Investigator — N.I. Pirogov National Medical and Surgical Center
Locations (1):
- N.I. Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slooter AJC, Otte WM, Devlin JW, Arora RC, Bleck TP, Claassen J, Duprey MS, Ely EW, Kaplan PW, Latronico N, Morandi A, Neufeld KJ, Sharshar T, MacLullich AMJ, Stevens RD. Updated nomenclature of delirium and acute encephalopathy: statement of ten Societies. Intensive Care Med. 2020 May;46(5):1020-1022. doi: 10.1007/s00134-019-05907-4. Epub 2020 Feb 13. No abstract available. PMID 32055887
- [Derived] Vinogradov OI, Ogarkova TK, Shamtieva KV, Alexandrov PV, Mushba AV, Kanshina DS, Yakovleva DV, Surma MA, Nikolaev IS, Gorst NK. Predictors of Acute Encephalopathy in Patients with COVID-19. J Clin Med. 2021 Oct 20;10(21):4821. doi: 10.3390/jcm10214821. PMID 34768339